CLINICAL TRIAL: NCT03189693
Title: Paravertebral Block for Postoperative Pain Management in Adult Patients Undergoing Appendectomy
Brief Title: Paravertebral Block for Pain Management After Appendectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Zoher Naja, Chairperson of Anesthesia and Pain Management Department, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 212006
Record Dates: First submitted 2017-06-13; First posted 2017-06-16 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Reduce Pain After Appendectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVB group (Experimental): Patients will receive two PVB injections at levels T12-L1 and L1-L2 using anesthetic mixture
  Interventions: Other: PVB; Other: GA; Other: Anesthetic injections
- Placebo (Placebo Comparator): Patients will receive two PVB injections containing placebo at levels T12-L1 and L1-L2
  Interventions: Other: Placebo; Other: GA

INTERVENTIONS:
Other: PVB — nerve stimulator-guided PVB will be performed at two levels
  Arms: PVB group
Other: Placebo — nerve stimulator-guided PVB containing placebo will be performed at two levels
  Arms: Placebo
Other: GA — All patients will receive general anesthesia.
Other: Anesthetic injections — 4 mL of the local anesthetic mixture is injected at each injection site. Each 20 mL of the local anaesthetic mixture contains: 8mL lidocaine 2%, 8 mL lidocaine 2% with epinephrine 5µg/mL and 4 mL bupivacaine 0.5%.
  Arms: PVB group

SUMMARY:
Paravertebral Block (PVB) was shown to be a successful and useful technique of anesthesia and analgesia. Its effect was evident in thoracic and abdominal surgeries. In the setting of appendectomy, somatic PVB has been used for pediatric patients. It was shown to decrease opioid consumption and provide prolonged pain relief. Hence, it would be beneficial to examine the analgesic effect of PVB on appendectomy in adult patients.

DETAILED DESCRIPTION:
Patients undergoing appendectomy will be randomly allocated into two equal groups using the sealed envelope technique. All patients will receive general anesthesia (GA). Patients in group I will receive two PVB injections at levels T12-L1 and L1-L2 using anesthetic mixture, while patients in Group II will receive placebo.

Paravertebral Block Technique Unilateral right side nerve stimulator-guided PVB is performed while patients are in the left lateral decubitis position. The appropriate levels for the PVB are determined by palpation of the spinous processes. An intervertebral line is drawn at the appropriate levels and the injection site is marked 2.5 cm lateral to the midline. After aseptic preparation of the skin, 1 mL 1% lidocaine is infiltrated at the injection sites. A 21-G nerve stimulation needle (Stimuplex; B. Braun, Melsungen, Germany) is advanced 1-2 cm perpendicularly to the skin using a nerve stimulating current of 2.5-5.0 mA, while closely watching for contractions of the abdominal muscles. The tip of the needle is adjusted to maintain muscle contractions while reducing the stimulating current to approximately 0.5-0.6 mA.

4 mL of the local anaesthetic mixture is injected at each injection site. Each 20 mL of the local anaesthetic mixture contains: 8mL lidocaine 2%, 8 mL lidocaine 2% with epinephrine 5µg/mL and 4 mL bupivacaine 0.5%.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Scheduled to undergo appendectomy

Exclusion Criteria:

* cardiac disease,
* developmental delay,
* neurologic deficit,
* allergies to any of the drugs routinely used in anesthesia management.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Analgesic consumption | 24 hours postoperatively
  The quantity of analgesics consumed will be recorded

SECONDARY OUTCOMES:
hemodynamic stability measured through mean arterial pressure (MAP). | Approximately 1 hour
  Intraoperative hemodynamic stability measured through mean arterial pressure (MAP)

CONTACTS AND LOCATIONS:
Locations (1):
- Makassed General Hospital, Beirut, Lebanon